CLINICAL TRIAL: NCT01730651
Title: A Phase II Study of High Dose Intensity Modulated Radiation Therapy in the Cervical Cancer With Metastatic Lymphadenopathies at Initial Diagnosis.
Brief Title: High Dose Intensity Modulated Radiation Therapy in the Cervical Cancer With Metastatic Lymphadenopathies.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Young Kim, PI, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS 12-615
Record Dates: First submitted 2012-10-15; First posted 2012-11-21 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Cervical Cancer
Keywords: cervical cancer with metastatic lymphadenopathies
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tomotherapy (Experimental): 1. Tomotherapy fraction size (Gy) = 0.4 x 진단 당시의 LN short diameter (cm) + 1.6 (pilot study range, 1.5-3.0 Gy)
  2. Total dose(summation dose with 3D-CRT) (Gy10) (EQD2, α/β=10 Gy) = 5 x 진단 당시의 LN short diameter (cm) + 56 (pilot study range, 54.6-78.0 Gy)
  Interventions: Radiation: Tomotherapy

INTERVENTIONS:
Radiation: Tomotherapy — IMRT boost of gross LNs
  1. Tomotherapy fraction size (Gy) = 0.4 x 진단 당시의 LN short diameter (cm) + 1.6 (pilot study range, 1.5-3.0 Gy)
  2. Total dose(summation dose with 3D-CRT) (Gy10) (EQD2, α/β=10 Gy) = 5 x 진단 당시의 LN short diameter (cm) + 56 (pilot study range, 54.6-78.0 Gy)

SUMMARY:
This phase II study of high dose intensity modulated radiation therapy in the cervical cancer with metastatic lymphadenopathies at initial diagnosis

DETAILED DESCRIPTION:
Lymph node (LN) involvement in cervical cancer is a poor prognostic factor(1). Although lymph node evaluation is not a part of the International Federation of Gynecology and Obstetrics (FIGO) staging system(2), it is generally performed as one of the initial workup of patients with cervical cancer by use of modern imaging tools for accurate evaluation of the disease extent and possible treatment adjustment. Kidd et al reported the positron emission tomography with [18F] fluorodeoxyglucose (FDG-PET)-positive lymph node rate is 47% at diagnosis in 560 patients. They also showed that within a stage, patients with PET-positive lymph nodes had significantly worse disease specific survival than those with PET-negative lymph nodes (p<0.001)(3).

Historically, dose escalation to the pelvic or para-aortic metastatic lymphadenopathies was not given as much attention as primary uterine cervical lesion partly because of the expected increased risk of bowel toxicity with when conventional radiotherapy technique was used. Unlike for the head and neck cancer where intensity modulated radiation therapy (IMRT) or tomotherapy was actively used for treatment of large lymphadenopathies and shown to produce improved disease control(4, 5) , there are few similar studies for cervical cancer. It is well known that more than 60 Gy10 2Gy equivalent dose (EQD2, α/β=10 Gy) is needed to control the gross tumor sized of 10 mm, containing 109 cells, according to the logarithmic cell killing(6). Theoretically, pelvic and para-aortic LNs (PAN) could not be controlled with the dose of 45-50 Gy10 EQD2, and we need to escalate the dose as much as possible with new radiation technology.

In the current is study, we evaluate the LNs control rate, toxicity rate, progression-free survival and overall survival in cervical cancer patients with lymphadenopathies and treated with high dose intensity modulated radiation therapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients (who have been adequately clinically staged) with primary, untreated, histologically confirmed carcinoma of the uterine cervix (including clear cell and small cell carcinoma), with metastatic lymphadenopathies (any of pelvis or PAN >1.5 cm in short diameter, with/without biopsy proven inguinal lymph node [ING])
2. Patients with Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, 2
3. Patients with adequate bone marrow function: absolute neutrophil count (ANC) greater than or equal to 1,500/mcl, platelets greater than or equal to 100,000/mcl at the beginning.
4. Patients with adequate renal function: creatinine equal to or less than 2.0 mg%.
5. Patients who have signed an approved informed consent and authorization

Exclusion Criteria:

1. Patients with recurrent LN(s) which was(were) previously irradiated.
2. Patients who have diagnosis of other malignance tumors except papillary or follicular thyroid cancer or skin cancer
3. Patients with metastatic lymphadenopathies other than pelvis, PAN, ING (e.g. supraclavicular or mediastinal metastatic lymphadenopathy)
4. Patients with distant organ metastasis (e.g. bone, lung, brain…)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2012-07-13 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | documented data of death, up to 3 years
  From date of initiation of radiotherapy until the date of documented date of death from any cause, assessed up to 3 years

SECONDARY OUTCOMES:
Disease-free survival (DFS) | documented date of progression or death, up to 3 years
  From date of initiation of radiotherapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  * Progression-free survival of lymph nodes(LNs) treated with high dose ② Regional LN (other than the LNs treated with high dose) failure-free survival ③ Distant organ (other than para-aortic LNs[PAN]) failure-free survival

OTHER OUTCOMES:
RTOG acute and late Toxicity | every follow-up date, up to 3 years
  ① Acute: gastrointestinal (GI), genitourinary (GU), bone marrow (BM)
  ② Late: GI, GU, lower extremity edema, treatment-related neuropathy, bone density change

CONTACTS AND LOCATIONS:
Overall Officials: Jooyoung Kim, M.D., Principal Investigator — National Cancer Center, Korea
Locations (2):
- South Korea (2):
  - National Cancer Center, Korea, Goyang-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: Undecided
undecided